CLINICAL TRIAL: NCT04273347
Title: Incidence of Neurogenic Paraosteoarthropathies (NPOA) in a Population of Brain Traumatized and Spinal Cord Injured Patients and Specific Markers of Early Neurogenic Paraosteoarthropathies Development"
Brief Title: Incidence of Neurogenic Paraosteoarthropathies in a Population of Brain Traumatized and Spinal Cord Injured Patients and Specific Markers of Early NPOA Development"
Acronym: BENTHOS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190623
Record Dates: First submitted 2019-11-22; First posted 2020-02-18 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Spinal Cord Injuries; Injury, Brain, Traumatic
MeSH Terms: conditions — Spinal Cord Injuries; Brain Injuries, Traumatic | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient with brain trauma: all patient with brain trauma in intensive care unit
  Interventions: Other: standard of care for patient with brain trauma and spinal cord injury
- patient with spinal cord injury: all patient with spinal cord injury in intensive care unit
  Interventions: Other: standard of care for patient with brain trauma and spinal cord injury

INTERVENTIONS:
Other: standard of care for patient with brain trauma and spinal cord injury — neurological examination, examination of articulation, infectious status, respiratory status, inflammatory status,kinesitherapy

SUMMARY:
Neurogenic paraosteoarthropathies are peri-articular bone formations that may occur as a result of central neurological injury. Their occurrence limits reeducation and recovery capacities. Neurogenic paraosteoarthropathies sometimes cause complications (pain, joint stiffness, vascular and nerve compression, pressure sores) in patients already suffering from severe neurological sequelae affecting functional prognosis. A lot of clinical research work has been carried out within Dr Salga team. Subsequently, a collaboration was born with fundamental research teams (Pr Levesque, Pr Le Bousse Kerdilès, Pr Banzet, Pr Genêt) allowing translational work between humans and animals. The clinical application of recent research findings now makes it possible to launch the very first prospective study on neurogenic paraosteoarthropathies.

DETAILED DESCRIPTION:
Based on the results of collaborative and translational (human-animal) work, investigators wish to conduct the first prospective study that would allow:

(i) To assess the incidence of Neurogenic paraosteoarthropathies (clinical suspicion and radiological confirmation). The prospective nature of this clinical data collection will make it possible to avoid the biases attributed to the retrospective studies conducted to date.

ii) Early detection of patients at risk of developing Neurogenic paraosteoarthropathies, using specific biomarkers and clinical parameters. Early diagnosis could prevent complications and functional impact of Neurogenic paraosteoarthropathies.

Investigators have chosen to restrict population to patients most at risk of developing Neurogenic paraosteoarthropathies as a result of the central neurological event in order to have 2 populations appear at the end of the study: a population with Neurogenic paraosteoarthropathies and a population without Neurogenic paraosteoarthropathies that can be compared.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female > 18 years old,
* brain trauma with initial Glasgow score < 8,
* or brain trauma with an initial Glasgow score between 8 and 14 associated with an Injury Severity Score (ISS) > 15 and surgery within 24 hours of admission or traumatic spinal cord injury with complete neurological impairment (initial para/tetraplegia),
* Complete traumatic spinal cord injury. Accident less than 48 hours old
* Informed consent signed by the patient or a family member

Exclusion Criteria:

* Age < 18 years,
* Hemorrhagic shock or blood transfusion greater than or equal to 4 red blood cells within 6 hours of the trauma (also include pre-hospital or first hospital red blood cells)
* Follow-up impossible over one year,
* Patient not living in the Paris region,
* Pregnant or breastfeeding woman,
* Patient under guardianship or curatorship,
* No affiliation to a social security scheme or universal mutual fund.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with brainTrauma or spinal cord injury upon arrival in intensive care
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Neurogenic Paraosteoarthropathies | 9 months
  Determine the incidence of Neurogenic Paraosteoarthropathies within 9 months of a brain trauma and/or spinal cord injury

SECONDARY OUTCOMES:
the incidence of Neurogenic Paraosteoarthropathies development within 9 months of a brain trauma | 9 months
  determine the incidence of Neurogenic Paraosteoarthropathies development within 9 months of a brain trauma
the incidence of Neurogenic Paraosteoarthropathies development within 9 months of a spinal cord injury, | 9 months
  determine the incidence of Neurogenic Paraosteoarthropathies development within 9 months of a spinal cord injury,
correlation between biological parameters from blood/plasma, urine and cerebrospinal fluid within 15 days of a central neurological injury and the occurrence of Neurogenic Paraosteoarthropathies within 9 months of the trauma | 15 days
  Determine if there is an correlation between biological parameters from blood/plasma, urine and cerebrospinal fluid within 15 days of a central neurological injury and the occurrence of POAN within 9 months of the trauma
a correlation between clinical parameters identified within 9 months of the neurological event and the occurrence of Neurogenic Paraosteoarthropathies within one year of the trauma, | 12 months
  Determine if there is a correlation between clinical parameters identified within 9 months of the neurological event and the occurrence of Neurogenic Paraosteoarthropathies within one year of the trauma,
a clinical-biological risk score for Neurogenic Paraosteoarthropathies within 9 months of the trauma | 9 months
  Create a clinical-biological risk score for Neurogenic Paraosteoarthropathies within 9 months of the trauma
the prognostic performance | 12 months
  Calculate the prognostic performance (of POAN occurrence in the year after the trauma) for the biological parameters statistically associated with Neurogenic Paraosteoarthropathies occurrence and for the risk score

CONTACTS AND LOCATIONS:
Overall Officials: Majorie Salga, MD, Principal Investigator — Hôpital Raymond Poincaré

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Torossian F, Guerton B, Anginot A, Alexander KA, Desterke C, Soave S, Tseng HW, Arouche N, Boutin L, Kulina I, Salga M, Jose B, Pettit AR, Clay D, Rochet N, Vlachos E, Genet G, Debaud C, Denormandie P, Genet F, Sims NA, Banzet S, Levesque JP, Lataillade JJ, Le Bousse-Kerdiles MC. Macrophage-derived oncostatin M contributes to human and mouse neurogenic heterotopic ossifications. JCI Insight. 2017 Nov 2;2(21):e96034. doi: 10.1172/jci.insight.96034. PMID 29093266
- [Result] Reznik JE, Biros E, Marshall R, Jelbart M, Milanese S, Gordon S, Galea MP. Prevalence and risk-factors of neurogenic heterotopic ossification in traumatic spinal cord and traumatic brain injured patients admitted to specialised units in Australia. J Musculoskelet Neuronal Interact. 2014 Mar;14(1):19-28. PMID 24583537